CLINICAL TRIAL: NCT06308692
Title: Molecular Diagnostics of Bacterial Infections and Antibiotic Resistance in Blood Samples and Rectal Swabs Using Real Time PCR-ARES PCR Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-11
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Drug Resistant Bacterial Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological samples (Other): Residual anonymized samples stored at -80°C at the Tropica Biobank of the DITM and for which diagnostic analysis for germ infection has previously been carried out at the DITM by blood culture and MDR surveillance in routine diagnostic rectal swab will be used.
  Interventions: Diagnostic Test: ARES PCR

INTERVENTIONS:
Diagnostic Test: ARES PCR — Real time PCR assays will be used for the identification of infecting microorganisms and the drug resistance they carry that allow their identification, such as KPC, VIM, IMP, NDM, Acinetobacter OXA, Oxa48, MCR.
  The validation of the method will be carried out in 100 (based on availability in Tropica Biobank) clinical samples: blood n=50 (positive, as for the negatives reference will be made to those already provided in the GENRES study) and rectal swabs ( positive n=40 and negative n=10) provided by the DITM. Sensitivity and specificity will be analyzed. As a reference for positivity and negativity data, reference will be made to routine diagnostic data obtained through standard operating procedures at the DITM laboratories.

SUMMARY:
Experimental study without drug and device, on pseudo-anonymized samples archived at the Tropica Biobank.

The objective is to evaluate the performance for the identification of microorganisms in blood samples and rectal swabs of real time PCR assays for the targets: KPC, VIM, IMP, NDM, Acinetobacter OXA, Oxa48, MCR.

The evaluations will be carried out taking into consideration the data obtained from the diagnostic routine at the DITM.

ELIGIBILITY:
Inclusion criteria:

* Samples of patients for whom blood culture and Multi Drug Resistant (MDR) surveillance tests were carried out in rectal swabs at the IRCCS Sacro Cuore Don Calabria Hospital
* Samples for which the Information and consent to the conservation of biological samples for research purposes at the Tropica Biobank has been signed

Exclusion criteria:

* Absence of data relating to positivity or negativity to the germs of interest
* Absence of stored residual material
* Absence of information and consent to the conservation of biological samples for signed research purposes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PCR results | Baseline
  Results (positive/negative and microorganism identification) obtained by real time PCR.

SECONDARY OUTCOMES:
Gene mutations | Baseline
  Results (resistant/susceptible) obtained by real time PCR in the identification of gene mutations that convey resistance to antibiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy